CLINICAL TRIAL: NCT06343220
Title: Project AWARE 2.0 to Improve Awareness, Willingness and Ability for Research and Enrollment in Clinical Research
Status: Completed | Type: Observational
Sponsor: Huntington Study Group (Network)
Collaborators: Roche Products Limited (Unknown); Neurotargeting LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: AWARE 2.0
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Huntington Disease
Keywords: HSG, HD, Observational
MeSH Terms: conditions — Huntington Disease; Charcot-Marie-Tooth Disease, Axonal, Type 2A2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Project AWARE 2.0 Survey is intended to gain knowledge about the feelings, attitudes, and beliefs of HD family members, care partners and others affected by HD towards the way drug trials and observational studies are communicated and conducted.

DETAILED DESCRIPTION:
The Project AWARE 2.0 Survey will be offered to HD families via HSG's online platform called myHDstory®. The survey will obtain input and knowledge about their feelings, attitudes, and beliefs concerning clinical research and the process by which HD studies are communicated and conducted. Project AWARE 2.0 is intended to provide the HD research community with the insight and tools to help (a) improve prospective research participants' awareness, willingness, and ability to participate in clinical research for HD; and (b) design clinical studies and trials in the future.

ELIGIBILITY:
Inclusion Criteria:

* Participants must either have HD or be at risk for having HD
* Participants must be 18 years of age or older
* Participants must live in the United States
* Inclusion of participants will not be based on race, gender, or ethnicity.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Must either have HD or be at risk for having HD.
Sampling Method: Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-12-22 (Actual); Study Completion 2025-12-22 (Actual)

PRIMARY OUTCOMES:
Examine awareness | December 2024
  To examine prospective research participants' awareness, willingness, and ability to participate in clinical research for HD.
Provide the HD research community with the insight. | December 2024
  Provide the HD research community with insight to design clinical studies and trials in the future.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Brown, MD, MS, Principal Investigator — HSG
Locations (1):
- Huntington Study Group, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The Project AWARE 2.0 Survey is intended to gain knowledge about the feelings, attitudes, and beliefs of HD family members, care partners and others affected by HD towards the way drug trials and observational studies are communicated and conducted. Answers to these questions will provide valuable information to the HD research community when designing and conducting drug trials and observational studies.
Time Frame: 2024